CLINICAL TRIAL: NCT03296098
Title: A Multi-center, Open-label, Non-comparative Study of the Safety and Contraceptive Efficacy of Continuous Daily Oral 10 mg of Ulipristal Acetate (UPA)
Brief Title: Study of the Safety and Efficacy of Ulipristal Acetate (UPA) Used Daily as a Contraceptive
Acronym: CCN013B
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn due to FDA feedback
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCN013B
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Contraception; Healthy Female
Keywords: Contraception; Healthy Female; Progestin; ulipristal acetate
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ulipristal acetate (Experimental): Subjects will be administered ulipristal acetate in 5 mg dosages and instructed to take two pills once daily for 6 months.
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate — Ulipristal aceteate 5 mg oral tablets to take two tablets daily.

SUMMARY:
This is a Phase IIb multicenter, open-label, non-comparative trial of continuous daily oral 10 mg of ulipristal acetate (UPA) to evaluate its contraceptive efficacy as the primary method of contraception.

DETAILED DESCRIPTION:
This is an open-label study being conducted at 18 centers. The dose of 10 mg was chosen for daily continuous use of ulipristal acetate (UPA). The study will enroll approximately 300 subjects to use the UPA for 6 months (182 days). In addition to contraceptive efficacy, safety, overall acceptability of the product, and the number of bleeding/spotting days will be assessed.

ELIGIBILITY:
Inclusion Criteria:

To enroll into the clinical trial, potential subjects must:

1. Be in good general overall health with no chronic medical conditions that result in periodic exacerbations that require significant medical care.
2. Be women between 18 and 35 years inclusive at the enrollment visit.
3. Have regular menstrual cycles that occur every 21-35 days when not using hormonal contraception.

   a. If subject is postpartum or post-abortal, she must have one menstrual bleed prior to enrollment.
4. Be seeking contraception, and willing to use the study drug as the only contraception method during their months of study participation.
5. If using a ring, patch, pill, or implant prior to study treatment, the subject must discontinue the active hormone at least 4 days, and no more than 7 days, prior to study drug initiation. Note that for combined oral contraceptive users, placebo pills are not counted as active hormone.
6. If using a hormonal intrauterine device (IUD) prior to study treatment, the IUD must be removed prior to study drug initiation; removal and study drug initiation can occur on the same day, but the subject must refrain from sexual intercourse for 7 days following IUD removal.
7. If using a copper IUD prior to study treatment, the IUD must be removed prior to study drug initiation; removal and study drug initiation can occur on the same day. The IUD removal and study drug initiation must occur during the first 7 days of a spontaneous menses.
8. If using a non-hormonal contraceptive method (e.g. condoms or withdrawal) prior to study treatment, drug initiation should occur within the first 7 days of a spontaneous menses.
9. If the woman has received a long-acting injectable contraceptive (e.g. depomedroxyprogesterone acetate) during the 10 months prior to screening, she must have resumed cyclic spontaneous menses (two menstrual bleeds) since last injection.
10. Have a negative urine pregnancy test at the enrollment visit.
11. Have an intact uterus and both ovaries.
12. In the opinion of the investigator, be willing and able to follow all study requirements, including use of the study product and be willing to record requested information on a daily diary.
13. Understand and sign an (Institutional Review Board) IRB approved informed consent form prior to screening activities (including fasting blood draws).
14. Have a diastolic blood pressure (BP) ≤95 mm Hg and systolic BP ≤145 mm Hg after 5 minutes in a sitting position at the enrollment visit. Hypertensive subjects who are treatment controlled and, in the judgment of the investigator, are good candidates require a waiver for participation.
15. Have a body mass index (BMI) < 40 kg/m2.
16. Be planning to have at least one act of heterosexual vaginal intercourse each month during study participation.
17. Be willing to accept an unknown risk of pregnancy during study participation.

Exclusion Criteria:

To enroll into the clinical trial, potential subjects must not:

1. Be women with irregular menstrual cycles defined as a variation in cycle length of more than 5 days.
2. Be planning pregnancy within their months of study participation.
3. Be currently breast-feeding or within 30 days of discontinuing breast feeding, unless the subject has already had a menses following discontinuation of breast feeding.
4. Have undiagnosed abnormal genital bleeding.
5. Have known hypersensitivity to the active substance UPA or any of the excipients of the study treatment.
6. Have a history of endometrial hyperplasia or malignancy.
7. Have abnormal Transvaginal Ultrasound (TVUS) or safety labs done at the screening visit recognized as clinically significant by the investigator (or medically qualified designee).
8. Have a previous history of endometrial ablation.
9. Have a previous history of liver disease or screening liver enzyme results more than three times the upper limit of normal values.
10. Have a known clinically significant Pap test abnormality, as managed by current local or national guidelines, that would require treatment during study participation.
11. Have any of the following known contraindication to progestin-only oral contraceptive (OC):

    1. History or existing breast cancer, or other hormone sensitive neoplasia;
    2. Current or history of ischemic heart disease or stroke while pregnant or taking birth control pills;
    3. Systemic Lupus Erythematosus with positive or unknown antiphospholipid antibodies;
    4. Benign or malignant liver tumors;
    5. Severe (decompensated) cirrhosis.
12. Have known or suspected alcoholism or drug abuse.
13. Have known HIV infection.
14. Have an anticipated need for regular condom use as defined as use of at least one condom per month after enrollment.
15. Have previously participated in the study.
16. Have a current need for exogenous hormones or therapeutic anticoagulants.
17. Have a current or history of deep vein thromboembolic disorder or aortic thromboembolism, including stroke and myocardial infarction
18. Have a current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive, unless she is stable on antidepressant medication.
19. Have concomitant use of medication thought to interact with UPA (per Summary of Product Characteristics (SPCs)) such as CYP3A4 inducers (rifampin, barbiturates, carbamazepine, bosentan, felbamate, griseofulvin, oxcarbazepine, phenytoin, St John's Wort, topiramate).
20. Have concomitant use of moderate or strong CYP3A4 inhibitors as identified by the FDA. Subjects who begin use of a moderate CYP3A4 inhibitor after study enrollment require a waiver to continue in the study.
21. Use any medications that can interfere with the metabolism of hormonal contraceptives, antibiotics that can interfere with metabolism of hormonal contraceptives, or any drugs designated by the FDA as falling in the Pregnancy and Lactation narrative subsections (formerly Category D or X medications).
22. Currently participate in any other trial of an investigational medicine or device or have participated in the three months before start of treatment or be planning to participate in another clinical trial during this study.
23. Have a history of a bariatric surgery procedure associated with malabsorption.
24. Be planning to undergo major surgery during study participation.
25. Live outside of the catchment area of the study site.
26. Have used UPA, including Ella, within 30 days prior to enrollment and not had a menses since using UPA.
27. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the contraceptive efficacy at 6 months based on the calculated Pearl Index for the evaluable for pregnancy population. | 6 months

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) during 6 month use of UPA. | 6 months
Changes from baseline in sodium levels (safety and tolerability). | 6 months
Changes from baseline in potassium levels (safety and tolerability). | 6 months
Changes from baseline in chloride levels (safety and tolerability). | 6 months
Changes from baseline in bicarbonate levels (safety and tolerability). | 6 months
Changes from baseline in fasting glucose levels (safety and tolerability). | 6 months
Changes from baseline in blood urea nitrogen levels (safety and tolerability). | 6 months
Changes from baseline in creatinine levels (safety and tolerability). | 6 months
Changes from baseline in calcium levels (safety and tolerability). | 6 months
Changes from baseline in total bilirubin levels (safety and tolerability). | 6 months
Changes from baseline in total alkaline phosphatase levels (safety and tolerability). | 6 months
Changes from baseline in total alanine aminotransferase levels (safety and tolerability). | 6 months
Changes from baseline in total aspartate transaminase levels (safety and tolerability). | 6 months
Changes from baseline in total albumin levels (safety and tolerability). | 6 months
Changes from baseline in total cholesterol levels (safety and tolerability). | 6 months
Changes from baseline in HDL cholesterol levels (safety and tolerability). | 6 months
Changes from baseline in LDL cholesterol levels (safety and tolerability). | 6 months
Changes from baseline in triglycerides levels (safety and tolerability). | 10 months
Changes from baseline in acceptability of UPA using an Acceptability Questionnaire (acceptability). | 6 months
Changes from baseline in bleeding pattern using a subject diary (tolerability). | 6 months
Changes from baseline in endometrial thickness using transvaginal ultrasound. | 6 months
Changes from baseline in endometrium using endometrial biopsy results. | 6 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Essential Access, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Hawaii, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - New York University, School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland MacDonald Women's Hospital, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Univeristy of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School (EVMS), Norfolk, Virginia